CLINICAL TRIAL: NCT00258713
Title: A 36-Week Extension to Protocol ISA04-03 to Evaluate the Safety and Efficacy of ISA247 in Patients With Plaque Psoriasis
Brief Title: A 36-Week Extension to Protocol ISA04-03
Acronym: SPIRIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aurinia Pharmaceuticals Inc. (Industry)
Responsible Party: Robert Huizinga, Isotechnika
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISA05-02
Record Dates: First submitted 2005-11-23; First posted 2005-11-28 (Estimated); Last update posted 2008-09-29 (Estimated); Status verified 2008-09

CONDITIONS: Psoriasis
Keywords: Randomized Controlled Trials; Immunosuppression; Adult; Chronic Disease; Dermatologic Agents; Female; Humans; Male; Middle Aged; Severity of Illness Index; Treatment Outcome; Quality of Life; Double-Blind Method
MeSH Terms: conditions — Psoriasis; Chronic Disease | interventions — voclosporin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator)
  Interventions: Drug: voclosporin
- 2 (Active Comparator)
  Interventions: Drug: voclosporin
- 3 (Active Comparator)
  Interventions: Drug: voclosporin

INTERVENTIONS:
Drug: voclosporin — voclosporin 0.2, 0.3, or 0.4 mg/kg BID

SUMMARY:
The purpose of this study is to determine the safety and efficacy of voclosporin in patients with plaque psoriasis.

DETAILED DESCRIPTION:
Psoriasis is a chronic skin condition that can have a significant impact on patient's physical and mental well being. The most common form of psoriasis is plaque psoriasis. Targeted treatments in psoriasis have been reported recently, yet cyclosporine, a calcineurin inhibitor (CNi) remains one of the treatments which has the greatest efficacy. Voclosporin represents the possibility of a calcineurin inhibitor which is not only as efficacious as cyclosporine A, but also has an improved toxicity profile.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-66 years inclusive at the time of visit 1.
* Diagnosed with plaque psoriasis ≥ 6 months.
* Currently participating in study ISA04-03 and completed the study up to and including Visit 9 of study ISA04-03.
* Not pregnant or nursing of planning to become pregnant during the course of the study
* Sexually-active women of child-bearing potential (including those who are < 1 year postmenopausal) and sexually-active men who are practicing a highly effective method of birth control. A highly effective method of birth control is defined as one that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly and will include implants, injectables, combined oral contraceptives, double-barrier method, sexual abstinence, or a sterile partner. Sexually-active men and women of child-bearing potential should continue to practice contraception as outlined above during treatment and for ≥ 3 months after the last dose of voclosporin.
* Written informed consent prior to any study related procedures.
* Able to keep study appointments and cooperate with all study requirements, in the opinion of the investigator.

Exclusion Criteria:

* Has generalized erythrodermic, guttate, or pustular psoriasis.
* Have other dermatoses that would interfere with the evaluation of psoriasis, at the discretion of the investigator.
* A current malignancy or history of malignancy within 5 years or a history of lymphoma at any time. Subjects can be enrolled with a history of squamous or basal cell carcinoma that has been surgically excised or removed with curettage and electrodesiccation.
* Has current, uncontrolled bacterial, viral, or fungal infection that requires intravenous antibiotics or antifungals.
* Has a current streptococcal infection that required oral antibiotics.
* A known history of tuberculosis.
* Serologic evidence or known latent human immunodeficiency virus (HIV), hepatitis B (HBV) or hepatitis C (HCV) virus.
* Uncontrolled hypertension as defined as 3 readings of systolic blood pressure ≥ 150 mm Hg or diastolic blood pressure ≥ 90 mm Hg.
* MDRD GFR ≤ 60 mL/min.
* Unstable renal function (variation in GFR ≥ 30%).
* Alanine transaminase, aspartate transaminase, or gamma-glutamyl transferase ≥ 3x upper limit of normal(ULN).
* White blood cell count ≤ 2.8x10 to the ninth power/L.
* Triglycerides ≥ 3x ULN.
* Is currently taking or requires the following prohibited medications or treatments during the treatment period: drugs potentiating the nephrotoxicity of voclosporin such as chronic NSAID's or ACE inhibitors, drugs interfering with it's pharmacokinetics; drugs considered to contribute to psoriasis flare; or, systemic and topical psoriasis medication (including psoralen/ultraviolet A light treatment) that may interfere with assessment of study drug efficacy.
* Has taken biological agent(s), except flu shots, tetanus shots, or boosters, within 3 months of the start of treatment. Biological agents include any virus, therapeutic serum, toxin, antitoxin, or analogous product applicable to the prevention, treatment, or cure of diseases or injuries of man.
* A history of clinically defined allergy to cyclosporine or any of the constituents of the voclosporin formulation (vitamin E, medium chain triglyceride oil, Tween 40, ethanol).
* A history of alcoholism or drug addiction within 1 year prior to study entry.
* Weighs < 45 kg (99 lbs) or > 140 kg (308 lbs).
* A history of disease, including mental/emotional disorder that would interfere with the subject's participation in the study, or that might cause the administration of ISA247 to pose a significant risk to the subject, in the opinion of the investigator.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2005-09; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
To investigate long-term safety and tolerability of voclosporin | Sixty weeks of continuous treatment

SECONDARY OUTCOMES:
To determine the proportion of subjects achieving and/or maintaining a PASI-75 | Sixty weeks of continuous treatment
To determine the proportion of subjects achieving and/or maintaining a reduction of 2 points in the SGA | Sixty weeks of continuous treatment
To evaluate the effect of voclosporin on subject quality of life | Sixty weeks of continuous treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, Principal Investigator — Innovaderm Research; Richard Langley, MD, FRCPC, Principal Investigator — Eastern Canada Cutaneous Research Associates Ltd.; Gilles Lauzon, PhD MD FRCPC, Principal Investigator — University of Alberta; Kim Papp, MD, PhD, Principal Investigator — Probity Medical Research; Neil Shear, MD, Principal Investigator — Ventana Clinical Research Corporation
Locations (23):
- Canada (23):
  - Isotechnika Investigational Site, Calgary, Alberta
  - Isotechnika Investigational Site, Edmonton, Alberta
  - Isotechnika Investigational Site, Vancouver, British Columbia
  - Isotechnika Investigational Site, Winnipeg, Manitoba
  - Isotechnika Investigational Site, Moncton, New Brunswick
  - Isotechnika Investigational Site, St. John's, Newfoundland and Labrador
  - Isotechnika Investigational Site, Halifax, Nova Scotia
  - Isotechnika Investigational Site, Barrie, Ontario
  - Isotechnika Investigational Site, Hamilton, Ontario
  - Isotechnika Investigational Site, London, Ontario
  - Isotechnika Investigational Site, Maple, Ontario
  - Isotechnika Investigational Site, Markham, Ontario
  - Isotechnika Investigational Site, Newmarket, Ontario
  - Isotechnika Investigational Site, North Bay, Ontario
  - Isotechnika Investigational Site, Oakville, Ontario
  - Isotechnika Investigational Site, Oshawa, Ontario
  - Isotechnika Investigational Site, Waterloo, Ontario
  - Isotechnika Investigational Site, Windsor, Ontario
  - Isotechnika Investigational Site, Laval, Quebec
  - Isotechnika Investigational Site, Montreal, Quebec
  - Isotechnika Investigational Site, Pointe-Claire, Quebec
  - Isotechnika Investigational Site, Saint Foy, Quebec
  - Isotechnika Investigational Site, Sherbrooke, Quebec

REFERENCES:
- [Background] Gregory CR, Kyles AE, Bernsteen L, Wagner GS, Tarantal AF, Christe KL, Brignolo L, Spinner A, Griffey SM, Paniagua RT, Hubble RW, Borie DC, Morris RE. Compared with cyclosporine, ISATX247 significantly prolongs renal-allograft survival in a nonhuman primate model. Transplantation. 2004 Sep 15;78(5):681-5. doi: 10.1097/01.tp.0000131950.75697.71. PMID 15371668
- [Background] Stalder M, Birsan T, Hubble RW, Paniagua RT, Morris RE. In vivo evaluation of the novel calcineurin inhibitor ISATX247 in non-human primates. J Heart Lung Transplant. 2003 Dec;22(12):1343-52. doi: 10.1016/s1053-2498(03)00033-0. PMID 14672749
- [Background] Abel MD, Aspeslet LJ, Freitag DG, Naicker S, Trepanier DJ, Kneteman NM, Foster RT, Yatscoff RW. ISATX247: a novel calcineurin inhibitor. J Heart Lung Transplant. 2001 Feb;20(2):161. doi: 10.1016/s1053-2498(00)00290-4. No abstract available. PMID 11250240